CLINICAL TRIAL: NCT00744367
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Effect of Taspoglutide on Glycemic Control Compared to Placebo in Patients With Type II Diabetes Mellitus Inadequately Controlled With Metformin Plus Pioglitazone
Brief Title: A Study of Taspoglutide Versus Placebo for the Treatment of Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin Plus Pioglitazone.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20963; 2008-001744-39
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone; taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Placebo in addition to continued stable metformin plus pioglitazone treatment. After the first 24 weeks patients on placebo will be switched to taspoglutide 10mg once weekly or taspoglutide 20mg once weekly (after 4 weeks of taspoglutide 10mg once weekly.
  Interventions: Drug: metformin; Drug: pioglitazone; Drug: placebo; Drug: taspoglutide
- Taspoglutide 10mg (Experimental): Taspoglutide 10mg once weekly in addition to continued stable metformin plus pioglitazone treatment
  Interventions: Drug: metformin; Drug: pioglitazone; Drug: taspoglutide
- Taspoglutide 10mg/20mg (Experimental): Taspoglutide 20 mg once weekly (after 4 weeks of taspoglutide 10 mg once weekly) in addition to continued stable metformin plus pioglitazone treatment.
  Interventions: Drug: metformin; Drug: pioglitazone; Drug: taspoglutide

INTERVENTIONS:
Drug: metformin — >1500 mg/day or maximum tolerated dose (MTD)
Drug: pioglitazone — >= 30 mg/day
Drug: placebo — sc once weekly
  Arms: Placebo
Drug: taspoglutide — 10 mg sc once weekly;
  Arms: Placebo; Taspoglutide 10mg
Drug: taspoglutide — 20 mg sc once weekly (after 4 weeks of taspoglutide 10 mg sc once weekly)
  Arms: Placebo; Taspoglutide 10mg/20mg

SUMMARY:
This 3 arm study will assess the efficacy of taspoglutide on glycemic control (as assessed by HbA1c) in patients with type 2 diabetes mellitus inadequately controlled with metformin plus pioglitazone, compared to placebo after 24 weeks of treatment. Patients will be randomized to one of 3 treatment arms: taspoglutide 10mg once weekly, taspoglutide 20 mg once weekly (after 4 weeks of taspoglutide 10 mg once weekly) or placebo, in addition to their continued stable metformin plus pioglitazone treatment. After the first 24 weeks patients on placebo will be switched to taspoglutide 10mg once weekly or taspoglutide 20mg once weekly (after 4 weeks of taspoglutide 10mg once weekly. The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years age;
* type 2 diabetes receiving pioglitazone (>= 30 mg/day) and metformin (>= 1500 mg/day) for at least 12 weeks prior to screening;
* HbA1c >=7.0% and <=10.0% at screening;
* BMI >= 25 (>23 for Asians) and <=45 kg/m2 at screening;
* stable weight +/-5% for at least 12 weeks prior to screening.

Exclusion Criteria:

* history of type 1 diabetes mellitus or acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma in the previous 6 months;
* evidence of clinically significant diabetic complications;
* clinically symptomatic gastrointestinal disease;
* myocardial infarction, coronary artery bypass surgery, post-transplantation cardiomyopathy or stroke within the previous 6 months;
* known hemoglobinopathy or chronic anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose; change from baseline in body weight; responder rates for HbA1c (target <=7.0%, <=6.5%); responder rates for body weight; beta cell function. | 24 weeks
Safety: adverse events, vital signs, physical examination, clinical laboratory tests, ECG and anti-taspoglutide antibodies. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (102):
- United States (71):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Buena Park, California
  - Lancaster, California
  - Loma Linda, California
  - Rancho Cucamonga, California
  - Roseville, California
  - San Diego, California
  - Walnut Creek, California
  - Wheat Ridge, Colorado
  - Hamden, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Chiefland, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Nampa, Idaho
  - Aurora, Illinois
  - Libertyville, Illinois
  - Evansville, Indiana
  - Des Moines, Iowa
  - Topeka, Kansas
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - New Orleans, Louisiana
  - Frederick, Maryland
  - Oxon Hill, Maryland
  - Detroit, Michigan
  - Ferndale, Michigan
  - Kalamazoo, Michigan
  - Biloxi, Mississippi
  - Olive Branch, Mississippi
  - City of Saint Peters, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albany, New York
  - Brooklyn, New York
  - Hudson, New York
  - Lake Success, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Mooresville, North Carolina
  - Wilmington, North Carolina
  - Bismarck, North Dakota
  - Athens, Ohio
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Norman, Oklahoma
  - Medford, Oregon
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Carlisle, Pennsylvania
  - Levittown, Pennsylvania
  - Melrose Park, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cranston, Rhode Island
  - Greer, South Carolina
  - Bellaire, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Federal Way, Washington
- Brazil (8):
  - Brasília
  - Forlateza
  - Fortaleza
  - Mogi Das Cruzes - Sp
  - Passo Fundo
  - Porto Alegre
  - Recife
  - São Paulo
- Canada (6):
  - Mount Pearl, Newfoundland and Labrador
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
- San José, Costa Rica
- France (4):
  - Bondy
  - Dijon
  - Nantes
  - Narbonne
- Germany (5):
  - Falkensee
  - Karlsruhe
  - Mainz
  - Neuwied
  - Potsdam
- Guatemala City, Guatemala
- Mexico (3):
  - Chihuahua City
  - Jalisco
  - Mexico City
- Puerto Rico (3):
  - Carolina
  - Guyanabo, San Juan
  - San Juan